CLINICAL TRIAL: NCT01909336
Title: Use of Isotonic Solutions Versus Hypotonic Solutions for Preventing Hospital Acquired Hyponatremia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Collaborators: Tecnologico de Monterrey (Other)
Responsible Party: Principal Investigator, Claudia Montserrat Flores Robles, MD, Claudia Montserrat Flores Robles, Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIvsSHnh
Record Dates: First submitted 2013-07-14; First posted 2013-07-26 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Sodium Chloride; Glucose; Hypotonic Solutions; Isotonic Solutions

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: 0.3% Saline in 3.3% dextrose (intravenous) (Active Comparator): Group 1: 0.3% Saline in 3.3% dextrose (intravenous)
  Interventions: Drug: 0.3% Saline in 3.3% dextrose
- Group 2: 0.45% Saline in 5% dextrose (intravenous) (Active Comparator): Group 2: 0.45% Saline in 5% dextrose (intravenous)
  Interventions: Drug: 0.45% Saline in 5% dextrose
- Group 3: 0.9% Saline in 5% dextrose (intravenous) (Active Comparator): Group 3: 0.9% Saline in 5% dextrose (intravenous)
  Interventions: Drug: 0.9% Saline in 5% dextrose

INTERVENTIONS:
Drug: 0.3% Saline in 3.3% dextrose — Hypotonic Solutions: 0.3% Saline in 3.3% dextrose
  Other Names: Hypotonic Solutions: 0.3% Saline + 3.3% dextrose
  Arms: Group 1: 0.3% Saline in 3.3% dextrose (intravenous)
Drug: 0.45% Saline in 5% dextrose — Hypotonic Solutions: 0.45% Saline in 5% dextrose
  Other Names: Hypotonic Solutions: 0.45% Saline in 5% dextrose
  Arms: Group 2: 0.45% Saline in 5% dextrose (intravenous)
Drug: 0.9% Saline in 5% dextrose — Isotonic Solutions 0.9% Saline in 5% dextrose
  Other Names: Isotonic Solutions 0.9% Saline in 5% dextrose
  Arms: Group 3: 0.9% Saline in 5% dextrose (intravenous)

SUMMARY:
The purpose of this study is to determine if isotonic solutions reduce the risk of hospital acquired hyponatremia compared with hypotonic solutions.

DETAILED DESCRIPTION:
Multicenter, Randomized, Controlled clinical trial.

The purpose of this study is to determine if isotonic solutions reduce the risk of hospital acquired hyponatremia compared with hypotonic solutions

This study will include 150 patients in 2 groups according to these type of pathology: group 1: medical conditions which includes respiratory problems (pneumonia, bronchiolitis, acute asthma attack) and acute gastrointestinal problems (bacterial or viral gastroenteritis) and group 2: surgical conditions (pre, peri or postoperative patients will be included). Each group will be randomized to receive 3 types of interventions: 0.3% Saline (hypotonic solution), 0.45% Saline (hypotonic solution) or 0.9% Saline (isotonic solution). In non-dehydrated patients the daily total volume of liquid infused will be determined by the volumetric Holliday- Segar* formula and the daily total volume will be calculated by adding the maintenance requirements (using the Holliday Segar formula) to the fluid deficit (according to percent of estimated weight**) in dehydrated patients.

The glucose concentrations in the first group will be 3.3%, and in group 2 and 3 will be 5%. The potassium concentration will be 20mEq/L in all groups. Blood samples will be collected before, 8 hours and 24 hours after the start of intravenous fluid, for the analysis of sodium, potassium, glucose, urea and creatinine. The adverse clinical outcomes at 8 and 24 hours of the start of intravenous fluid will also be recorded. The sodium plasma level, the incidence of hyponatremia and the adverse clinical outcomes will be compared.

*0-10 kilogram (kg): 100ml/kg per day; 10-20 kg: 1000 ml + 50 ml/kg/day over 10 kg; >20 kg: 1500 ml + 20ml/ kg over 20kg

** In patients under 10 kg correspond to a loss of 5% (50 mL/kg) in mild dehydration and 10% in moderate dehydration. In 10 kg or more: 3% (30 mL/kg) in mild dehydration and 6% (60 mL/kg) in moderate dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 months to 15 years.
* Need for intravenous fluids for 8 hours or more.
* Normal serum sodium at the beginning of the study of the study (135-145 mEQ/L).
* Acute respiratory problems (acute asthma attack, bronchiolitis or pneumonia).
* Acute gastrointestinal disorders (viral o bacterial gastroenteritis).
* Elective surgical procedures.
* Pre, peri o post operative patients (acute appendicitis, intussusception, intestinal perforation, ileus).

Exclusion Criteria:

* Severe hyponatremia (serum sodium < 125 mEq/L).
* Severe hypernatremia (serum sodium >155 mEq/L).
* Need for intravenous fluids for less than 8 hours according with their treating physician.
* Severe dehydration or Shock.
* Preexisting chronic diseases (renal diseases, heart diseases or endocrine disorders).
* Neurologic diseases.
* Head trauma.
* Cerebral edema or Intracranial hypertension.
* Diabetic ketoacidosis.
* Use of diuretics one week or less before the study.
* Need for admission to the pediatric critical intensive care unit

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Montserrat Flores Robles, MD, Principal Investigator — Tecnologico de Monterrey; Carlos Alberto Cuello García, MD, Study Director — Centro de Medicina Basada en Evidencias, Escuela de Medicina y Ciencias de la Salud, Tecnológico de Monterrey.

REFERENCES:
- [Background] Moritz ML, Ayus JC. Hospital-acquired hyponatremia--why are hypotonic parenteral fluids still being used? Nat Clin Pract Nephrol. 2007 Jul;3(7):374-82. doi: 10.1038/ncpneph0526. PMID 17592470
- [Background] Choong K, Kho ME, Menon K, Bohn D. Hypotonic versus isotonic saline in hospitalised children: a systematic review. Arch Dis Child. 2006 Oct;91(10):828-35. doi: 10.1136/adc.2005.088690. Epub 2006 Jun 5. PMID 16754657
- [Background] Montanana PA, Modesto i Alapont V, Ocon AP, Lopez PO, Lopez Prats JL, Toledo Parreno JD. The use of isotonic fluid as maintenance therapy prevents iatrogenic hyponatremia in pediatrics: a randomized, controlled open study. Pediatr Crit Care Med. 2008 Nov;9(6):589-97. doi: 10.1097/PCC.0b013e31818d3192. PMID 18838929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in the paediatric and emer- gency departments of the Hospital Regional Materno Infantil de Alta Especialidad in Nuevo Leon, Mexico between August 2013 and February 2014.
Groups:
- Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous): Group 1: 0.3% Saline in 3.3% dextrose (intravenous): Hypotonic Solutions
- Group 2: 0.45% Saline in 5% Dextrose (Intravenous): Group 2: 0.45% Saline in 5% dextrose (intravenous): Hypotonic Solutions
- Group 3: 0.9% Saline in 5% Dextrose (Intravenous): Group 3: 0.9% Saline in 5% dextrose (intravenous): Isotonic Solutions
Period: Overall Study
Arm/Group | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous)
Started | 53 | 53 | 55
Completed | 49 | 50 | 52
Not Completed | 4 | 3 | 3
Not completed — Lost to Follow-up | 4 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous) | Total
Number analyzed (Participants) | 49 | 50 | 52 | 151
Age, Continuous [Mean (Standard Deviation); unit: months] | 63.5 (56.1) | 54.6 (55.9) | 58.8 (57.7) | 58.9 (56.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 25 | 66
  Male | 28 | 30 | 27 | 85
Dehydration (mild), n [Number; unit: participants] — Dry mucous membranes in association with normal hemodynamic measurements
  participants | 10 | 13 | 10 | 33
Systolic blood pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 101.1 (11.2) | 99.4 (9) | 99.8 (11.4) | 100.1 (10.5)
Heart rate, bpm [Mean (Standard Deviation); unit: bpm] | 124 (25) | 126 (29) | 128 (28) | 126 (27)
Serum sodium, mmol/L [Mean (Standard Deviation); unit: mmol/L] | 135 (2.8) | 135.8 (3.1) | 135.8 (3.2) | 135.5 (3)
Serum osmolarity, mOsm/L [Mean (Standard Deviation); unit: mOsm/L] | 277.4 (10.6) | 278 (16.2) | 281.4 (9.5) | 279 (8.6)
Normonatremic, n [Number; unit: participants] — defined as serum sodium 135-145 mmol/L
  participants | 30 | 34 | 34 | 98
Hyponatraemia, n [Number; unit: participants] — defined as serum sodium < 135 mmol/L.
  participants | 19 | 16 | 16 | 51
Hypernatremic, n [Number; unit: participants] — defined as serum sodium > 145 mmol/L.
  participants | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Hospital Acquired Hyponatremia
Description: Serum sodium less than 135 mEq/L at 8 hours in a patient with normal serum sodium (135 mEq/L to 145mEq/L) at the beginning of the study
Time Frame: 8 hours
Measure: Number; unit: participants
Arm/Group | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous)
Number analyzed (Participants) | 30 | 34 | 34
participants | 10 | 11 | 1

2. Secondary Outcome: Dysnatraemias at T8
Description: hyponatraemia (defined as serum sodium < 135 mmol/L), normonatremia (defined as serum sodium 135-145 mmol/L) or hypernatraemia (defined as serum sodium > 145 mmol/L)
Time Frame: 8 hours
Measure: Number; unit: participants
Arm/Group | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous)
Number analyzed (Participants) | 49 | 50 | 52
participants
  Normonatremia | 26 | 30 | 47
  Hyponatremia | 23 | 20 | 3
  Hypernatremia | 0 | 0 | 2

3. Secondary Outcome: Adverse Reactions Attributed to Acute Plasma Sodium Changes
Description: Adjudicated Morbidity Attributed to Acute Plasma Sodium Changes assessed at 8 hours
Time Frame: 8 hours
Measure: Number; unit: Minor Adverse Reactions
Arm/Group | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous)
Number analyzed (Participants) | 49 | 50 | 52
Minor Adverse Reactions | 12 | 13 | 11

ADVERSE EVENTS:
Arm/Group | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous)
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 12/49 | 13/50 | 11/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 0.3% Saline in 3.3% Dextrose (Intravenous) (N=49) | Group 2: 0.45% Saline in 5% Dextrose (Intravenous) (N=50) | Group 3: 0.9% Saline in 5% Dextrose (Intravenous) (N=52)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3)
Fever (General disorders) | 4 (4) | 9 (9) | 4 (4)
Drowsiness (General disorders) | 2 (2) | 0 (0) | 2 (2)
Dehydration (General disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No